CLINICAL TRIAL: NCT06820866
Title: Non-invasive Diagnosis of Idiopathic Nephrotic Syndromes : DNI-SNI
Brief Title: Non-invasive Diagnosis of Idiopathic Nephrotic Syndromes
Acronym: DNI-SNI
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP241612; 2024-A02829-38 (Other: IDRCB number)
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Idiopathic Nephrotic Syndrome (INS)
Keywords: Kidney disease; Creatinine; DNI-SNI; Renal disease; Nephrotic Syndromes; Renal biopsy; Diagnostic score; Idiopathic Nephrotic Syndromes
MeSH Terms: conditions — Nephrosis, Lipoid; Kidney Diseases; Nephrotic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Renal biopsy (RB) is the reference diagnostic procedure for Idiopathic Nephrotic Syndrome (INS). It is an invasive procedure, particularly risky during the acute phase of nephrotic syndrome when anticoagulation therapy is required.

By identifying serum antibodies that allow for the non-invasive diagnosis of the main differential diagnoses of INS, (Membranous Nephropathy), the development of a non-invasive diagnostic tool for INS could help reduce the morbidity associated with the invasive renal biopsy procedure, minimizing the risk of incorrect diagnosis. We developed a diagnostic score, the SNIT, from routine clinical and biological variables to allow INS diagnoses in patients for whom detection of blood antibodies of Membranous Nephropathy were negative. The main goal of this study is to validate this diagnosis score in a prospective study, to allow INS diagnosis without renal biopsy.

DETAILED DESCRIPTION:
Medical management will not be altered by the protocol, and patients will be treated according to the practices of each center.

The investigator will offer participation in the study to all eligible consecutive patients in their center. They will provide an information sheet and answer any questions the patient may have. After obtaining the patient's non-opposition, the following clinical and biological data will be collected:

(Age, sex, medical and surgical history, BMI at admission, systolic and diastolic blood pressure at admission, presence of lower limb edema, CBC, blood electrolyte levels, urea, creatinine, albumin levels, urinary electrolytes, proteinuria, albuminuria, urine culture, antinuclear antibodies, serum protein electrophoresis, serum protein immunofixation, complement fractions C3 and C4, lipid profile).

The SNIT calculation will be performed automatically in the CRF from the variables it comprises, but will not be visible to the investigator.

As part of patient care, patients will be followed up one month after inclusion. During this visit, the evolving biological data (creatinine, albumin levels, proteinuria, albuminuria) and the treatment administered will be collected from the patient's medical records.

The final diagnosis will be collected as soon as it is available (within a maximum of 4 months for the completion and reporting of the histopathological results). Histological data will be collected from the report of the pathologist who examined the renal biopsy (available in the medical record). (In the case of INS: presence or absence of segmental and focal hyalinosis lesions, percentage of fibrosis).

The objectives of this study will be :

1. Evaluate the diagnostic performance of SNIT compared to renal biopsy (reference examination) for the diagnosis of Idiopathic Nephrotic Syndrome (INS)
2. Evaluate the other diagnostic parameters of the SNIT test.
3. Evaluate the avoidable costs
4. Evaluate the theoretical risks of a misdiagnosis of INS (through diagnostic delay and its consequences, as well as the risk of unnecessary corticosteroid treatment).

Duration of participant involvement and study duration:

The inclusion period will be 24 months. The follow-up period for participants will be a maximum of 4 months (until the histological diagnosis is returned). Therefore, the total duration of the research will be a maximum of 28 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Hospitalized for a first episode of nephrotic syndrome (proteinuria greater than 3g/g and albumin level < 30g/L)
* Negative anti-PLA2r antibodies in the blood
* Requirement for a renal biopsy for diagnostic purposes

Exclusion Criteria:

* Patients with known lupus nephropathy (prior to the current episode)
* Patients with known IgA nephropathy (prior to the current episode)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The diagnostic management of pediatric nephrotic syndrome is already covered by specific guidelines.
  Therefore, the population of our study will consist of adults over 18 years of age presenting with a first episode of nephrotic syndrome, without detectable anti-PLA2r antibodies in the serum (since their presence indicates the diagnosis of MN), and for whom a renal biopsy is indicated and performed for diagnostic purposes
Sampling Method: Non-Probability Sample
Enrollment: 265 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity of the SNIT score (threshold = 0.36) and their 95% confidence interval | 4 months

SECONDARY OUTCOMES:
Proportion of biopsies avoided with the use of SNIT. Proportions of diagnostic errors. Negative and positive predictive values and likelihood ratios of SNIT. | 4 months
Avoidable costs: costs of biopsies, impact on nephrology services. | 4 months
Estimation of the number of hospitalization days with the use of SNIT, and comparison with the actual number of hospitalization days. | 4 months
  The theoretical number of hospitalization days with the use of SNIT (i.e., estimated from the CRH data, subtracting the days of hospitalization required for renal biopsy in the case of a positive test).
  Adverse effects of corticosteroid treatment: infections, edema syndrome, corticosteroid-induced diabetes, heart failure decompensation.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre LAHENS, Dr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Néphrologie et Dialyses, Hôpital Tenon, Paris, France, France

IPD SHARING:
Plan to Share IPD: No